CLINICAL TRIAL: NCT06172478
Title: HERTHENA-PanTumor01 (U31402-277): A Phase 2, Multicenter, Multicohort, Open-Label, Proof of Concept Study of Patritumab Deruxtecan (HER3-DXd; U3-1402) in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of HER3-DXd in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U31402-277; 2023-507641-29-00 (Other: EU CTIS); jRCT2031230575 (Other: jRCT)
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Melanoma; Head and Neck Cancer; Gastric Cancer; Ovarian Carcinoma; Cervical Cancer; Endometrial Cancer; Bladder Cancer; Esophageal Cancer; Pancreatic Carcinoma; Prostate Cancer; Non-small Cell Lung Cancer (NSCLC); Lung Cancer; Breast Cancer
Keywords: Advanced Solid Tumor; Melanoma; Head and Neck Cancer; Gastric Cancer; Ovarian carcinoma; Cervical cancer; Endometrial cancer; Bladder cancer; Esophageal carcinoma; Pancreatic carcinoma; Prostate cancer; Patritumab Deruxtecan; HER3-DXd; U3-1402; Lung Cancer; Breast Cancer
MeSH Terms: conditions — Melanoma; Head and Neck Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Breast Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HER3-DXd Monotherapy (Experimental): Participants with locally advanced unresectable or metastatic cancer (melanoma, head and neck, gastric cancer, ovarian carcinoma, cervical cancer, endometrial cancer, bladder cancer, esophageal carcinoma, pancreatic carcinoma, prostate cancer, second-line gastric cancer, lung cancer, and breast cancer) will receive an intravenous infusion of HER3-DXd monotherapy 5.6 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: HER3-DXd

INTERVENTIONS:
Drug: HER3-DXd — Intravenous infusion 5.6 mg/kg administered Q3W on Day 1 of each 21-day cycle
  Other Names: Patritumab Deruxtecan; U3-1402

SUMMARY:
This is a proof-of-concept study designed to investigate HER3-DXd monotherapy in locally advanced unresectable or metastatic solid tumors. The study is enrolling cohorts of participants with melanoma [cutaneous/acral], squamous cell carcinomas of the head and neck (SCCHN), HER2-negative gastric cancer ovarian carcinoma, cervical cancer, endometrial cancer, bladder cancer, esophageal carcinoma, pancreatic carcinoma, prostate cancer, second-line gastric cancer, lung cancer, and breast cancer.

DETAILED DESCRIPTION:
This study is designed to assess the safety and efficacy of HER3-DXd monotherapy in subjects with refractory locally advanced unresectable or metastatic solid tumors who have been previously treated with ≥1 prior line of systemic anticancer therapy.

The primary objective of the study is to assess the efficacy of HER3-DXd monotherapy for each type of indicated locally advanced unresectable or metastatic tumor. Secondary objectives include the assessment of safety and tolerability, efficacy, and pharmacokinetics of HER3-DXd monotherapy for each type of indicated locally advanced unresectable or metastatic tumor. HER3 protein expression in tumor tissue and its relationship with HER3-DXd efficacy will also be evaluated.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be eligible for enrollment into the study:

1. Sign and date the informed consent form prior to the start of any study-specific qualification procedures. A separate tissue screening consent will be obtained from all subjects to meet the baseline tumor tissue requirement.
2. Participants aged ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years old).
3. Has locally advanced unresectable or metastatic disease (not curable by surgery or radiation) as follows:

   Cutaneous (acral and non-acral) melanoma
   1. Histologically or cytologically confirmed cutaneous (acral or non-acral) melanoma
   2. Disease progression while on or after having received treatment with ≥1 prior line of anti-programmed cell death protein (PD-1) or anti-programmed death-ligand 1 (PD-L1) based therapy (previous use of other immune checkpoint inhibitors [ICIs] [ie, anti-CTLA4, anti- LAG-3] is acceptable). Prior anti-PD-(L)1 therapy in the adjuvant setting is allowed if there is recurrence within 12 weeks of the last dose. If the participant had BRAFm melanoma, they must have had disease progression on BRAF/MEK inhibitor therapy as well.

      Squamous cell carcinomas of the head and neck
   3. Squamous cell carcinoma of the head and neck (with a primary location of oral cavity,oropharynx, larynx, hypopharynx) that is human papillomavirus (HPV) positive or negative (as determined by local standard). Excludes tumor location in the nasopharynx, nasal cavity, paranasal sinuses, and unknown primary locations.
   4. Disease progression after having received treatment with ≥1 and <3 prior lines of systemic therapy in the unresectable recurrent or metastatic setting.

      Must have had disease progression on anti-PD-(L)1 (either as monotherapy or in combination with chemotherapy or other therapies). Must also have had disease progression on a platinum-based chemotherapy (PBC) regimen either in the recurrent or metastatic setting or in the locally advanced setting with curative intent.

      Gastric or GEJ adenocarcinoma
   5. Tumor tissue must be confirmed as negative for HER2 expression (immunohistochemistry [IHC] 0/1+ or IHC 2+/in situ hybridization negative) as classified by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines and determined prior to enrollment by assessment in a local laboratory that is Clinical Laboratory Improvement Amendments certified (US sites) or accredited based on specific country regulations.
   6. Disease progression after having received treatment with ≥2 prior lines of therapy that include PBC with or without anti-PD-1 therapy.

      Ovarian Carcinoma
   7. Pathologically documented high-grade serous epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
   8. Documented disease progression ≥4 weeks after the last dose of PBC and <6 months of last dose of PBC in the advanced or metastatic setting. Prior use of folate reductase alpha targeting antibody-drug conjugate (ADC) (ie, mirvetuximab soravtansine) is allowed.

      Cervical Cancer
   9. Pathologically or cytologically documented recurrent or persistent squamous, adenosquamous, or adenocarcinoma of the uterine cervix.
   10. Disease progression after having received ≥1 line of systemic therapy in the recurrent or metastatic setting. This may include prior anti-PD-(L)1 treatment and/or tissue factor directed ADC (tisotumab vedotin [TV]) per regional standard of care.

       Endometrial Cancer
   11. Pathologically or cytologically documented endometrial cancer (carcinoma of any histological sub-type or endometrial carcinosarcoma), irrespective of microsatellite instability (MSI) or mismatch repair (MMR) status.
   12. Documented disease progression after having received ≥1 prior line of therapy (maximum of 3) PBC containing systemic treatment and an anti-PD(L)-1 therapy-containing regimen (combined or sequential) in the advanced/metastatic setting.

       Bladder Cancer
   13. Pathologically or cytologically documented locally advanced/unresectable or metastatic urothelial carcinoma of the bladder, renal pelvis, ureter, or urethra. Histological variants are allowed if urothelial histology is predominant. Small cell/neuroendocrine tumors are not allowed even if mixed histology.
   14. Relapsed or progressed after treatment with ≥1 prior line of therapy (maximum of 3) that contains anti-PD-(L)1 therapy in the perioperative or metastatic setting. At least 1 line of therapy must also contain one of the following treatment modalities: chemotherapy or enfortumab vedotin. Prior fibroblast growth factor receptor (FGFR)-inhibitor treatment for those who are eligible are allowed.

       * Required treatments can be given in combination or sequentially
       * Prior cisplatin-based therapy or PD-(L)1 inhibitor therapy given for the treatment of muscle invasive urothelial carcinoma is counted as 1 line of therapy
       * The same regimen administered twice in different disease settings will be counted as 1 line of prior therapy
       * Participants in the second-line setting who have previously received enfortumab vedotin and pembrolizumab in combination can be enrolled.

       Esophageal Carcinoma
   15. Pathologically or cytologically documented esophageal squamous cell carcinoma.
   16. Must have documented disease progression after having received 2 prior lines of therapy including previous PBC with or without an anti-PD-1 therapy-containing regimen (combined or sequential) in the advanced/metastatic setting.

       Pancreatic Carcinoma
   17. Pathologically or cytologically documented unresectable or metastatic pancreatic adenocarcinoma.
   18. Relapsed or disease progression after having received 1 prior line of systemic therapy in the locally advanced/metastatic setting.

       Prostate Cancer
   19. Pathologically or cytologically documented unresectable locally advanced or metastatic castration-resistant prostate cancer (CRPC).
   20. Adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology.
   21. Surgically or medically castrated, with testosterone levels of <50 ng/dL.
   22. Documented objective progression as determined by radiographic progression for subjects with measurable disease after androgen deprivation.
   23. Relapsed or disease progression after having received treatment with ≥1 of the following novel hormonal agents: abiraterone, enzalutamide, apalutamide, or darolutamide.
   24. Relapsed or disease progression after having received ≥1 cytotoxic chemotherapy regimen that included a taxane.

       Gastric Cancer 2L
   25. Must have had gastric or GEJ adenocarcinoma confirmed as negative for HER2 expression (IHC 0/1+ or IHC 2+/in situ hybridization negative) as classified by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines and determined prior to enrollment by assessment in a local laboratory that is Clinical Laboratory Improvement Amendments certified (US sites) or accredited based on specific country regulations.
   26. Disease progression after having received treatment with only 1 prior line of systemic anti-cancer therapy that includes 5-FU-based chemotherapy with or without an anti-PD-1 therapy. For subjects whose tumors are claudin (CLDN) 18.2 positive, treatment with 5-FU based chemotherapy with CLDN18.2 directed therapy in the first-line setting is allowed.

   Non-small Cell Lung Cancer aa. Histologically or cytologically documented metastatic or locally advanced nonsquamous NSCLC not amenable to curative surgery or radiation bb. Documentation of absence of actionable driver mutation (ie, ALK rearrangement, BRAF V600E mutation, EGFR-activating mutations [exon 19 deletion or L858R mutation], EGFR exon 20 insertion mutation, HER2 mutation, KRAS G12C mutation, MET exon 14 skipping mutation, NTRK 1/2/3 gene fusion, RET rearrangement, or ROS1 rearrangement). New testing for these genomic alterations is not required for Screening.

   cc. Relapsed or disease progression after receiving only anti-PD-(L)1 and PBC (ie, platinum doublet) administered in combination or sequentially for metastatic disease.

   Breast Cancer dd. Pathologically documented breast cancer that is assessed as HER2 negative (IHC2+/ISH-, IHC1+, or IHC0 per ASCO/CAP guidelines), and HR positive (either ER and/or PgR positive [ER or PgR ≥1%] per ASCO/CAP guidelines). The HER2 and HR results must be from a tumor sample obtained in the metastatic setting.

   ee. Participant must have received one line of chemotherapy for mBC, but not more than one line and must have a clinically or radiologically documented evidence of tumor progression on or after CDK 4/6 inhibitor combined with endocrine therapy; previous treatments with phosphoinositide 3-kinase (PI3K) inhibitors, mammalian target of rapamycin (mTOR) inhibitors, protein kinase B (PKB) inhibitors also known as AKT-inhibitors and poly ADP ribose polymerase (PARP)-inhibitors are allowed.
4. Has ≥1 measurable lesion on CT or MRI as per RECIST v1.1 by investigator assessment. Prostate cancer participants with bone only disease may be eligible.
5. Provides a pretreatment tumor tissue sample that meets 1 of the following collection requirements:

   1. Tumor biopsy from ≥1 lesion not previously irradiated and performed since progression with the most recent systemic cancer therapy regimen and prior to signature of the tissue ICF (ARCHIVAL PRETREATMENT sample).

      OR
   2. Newly obtained pretreatment tumor biopsy from ≥1 lesion not previously irradiated and amenable to sampling, after signature of tissue ICF (FRESH PRETREATMENT sample)
6. Has Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at screening.

Exclusion Criteria

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Has HER2-positive gastric cancer as classified by ASCO-CAP guidelines and determined prior to enrollment by assessment in a local laboratory that is Clinical Laboratory Improvement Amendments certified (US sites) or accredited based on specific country regulations.
2. Has nasopharyngeal cancer.
3. Has mucosal or uveal melanoma.
4. Has a history of (non-infectious) interstitial lung disease (ILD), that required corticosteroids, has current ILD/pneumonitis, or suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
5. Has clinically severe respiratory compromise (based on the investigator's assessment) resulting from intercurrent pulmonary illnesses
6. Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone daily or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to Cycle 1 Day 1.

   Participants who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study.
7. Had prior treatment with an anti-HER3 antibody and/or antibody-drug conjugate (ADC) that consists of an exatecan derivative that is a topoisomerase I inhibitor (eg, trastuzumab deruxtecan).
8. Has history of other active malignancy within 3 years prior to Cycle 1 Day 1, except the following:

   1. Adequately treated nonmelanoma skin cancer
   2. Adequately treated intraepithelial carcinoma of the cervix
   3. Any other curatively treated in situ disease
9. Has any evidence of severe or uncontrolled diseases (eg, active bleeding diatheses, active serious infection) psychiatric illness/social situations, geographical factors, substance abuse, or other factors that, in the investigator's opinion, make it high risk for the subject to participate in the study or that would jeopardize compliance with the protocol
10. Has previously received topoisomerase-1 inhibitors (e.g., irinotecan) treatment in the advanced or metastatic disease setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Objective Response Rate Assessed by Investigator Following HER3-DXd Monotherapy (All Cohorts Except Prostate Cancer Cohort) | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 27 months
  Confirmed objective response rate (ORR) is defined as the sum of the complete response (CR) rate and partial response (PR) rate based on investigator by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Proportion of Participants Achieving a ≥50% Decrease in PSA (Prostate Cancer Cohort Only) | Baseline, each cycle before infusion (each cycle is 21 days), and end of treatment, up to approximately 27 months

SECONDARY OUTCOMES:
Overall Number of Participants With Treatment-emergent Adverse Events Following HER3-DXd Monotherapy (All Cohorts) | Baseline up to 27 months
  Adverse events (AEs) will be coded using MedDRA and AEs and will be graded by using NCI-CTCAE v5.0.
Duration of Response As Assessed by Investigator Following HER3-DXd Monotherapy (All Cohorts Except Prostate Cancer Cohort) | From the date of first documentation of confirmed response (CR or PR) to the first documentation of objective progression or to death due to any cause, whichever occurs first, up to approximately 27 months
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first documentation of progressive disease (PD) or death. The DoR will be calculated for responding participants (PR or CR) only.
Clinical Benefit Rate As Assessed by Investigator Following HER3-DXd Monotherapy (All Cohorts Except Prostate Cancer Cohort) | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 27 months
  Clinical benefit rate (CBR) is the proportion of participants with a best overall response of confirmed CR, confirmed PR, or SD lasting ≥183 days.
Disease Control Rate As Assessed by Investigator Following HER3-DXd Monotherapy (All Cohorts Except Prostate Cancer Cohort) | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 27 months
  Disease control rate is defined as the proportion of participants who have achieved a best overall response of confirmed CR, confirmed PR, or SD (or non-CR/non-PD) by investigator assessment per RECIST v1.1.
Time to Response As Assessed by Investigator Following HER3-DXd Monotherapy (All Cohorts Except Prostate Cancer Cohort) | From the start date of study drug to the date of the first documentation of response (CR or PR) that is subsequently confirmed, up to approximately 27 months
  Time to response (TTR) will be calculated for confirmed responders only.
Progression-free Survival As Assessed by Investigator Following HER3-DXd Monotherapy (All Cohorts Except Prostate Cancer Cohort) | From the start date of study drug to the earlier date of the first objective documentation of radiographic disease progression as assessed by investigator per RECIST v1.1 or death due to any cause, whichever occurs first, up to approximately 27 months
Overall Survival Following HER3-DXd Monotherapy (All Cohorts) | From the start date of study drug to the date of death due to any cause, whichever occurs first, up to approximately 27 months
Pharmacokinetic Parameter Maximum Serum Concentration for HER3-DXd (All Cohorts) | Cycles 1-4, 6, 8: Day 1, predose and postdose; Cycles 1 and 3: Day 1, 2 hours and 4 hours postdose; Cycles 1 and 3: Day 8, Day 15 (each cycle is 21 days)
  Maximum serum concentration (Cmax) will be assessed using non-compartmental methods.
Pharmacokinetic Parameter Time to Maximum Serum Concentration for HER3-DXd (All Cohorts) | Cycles 1-4, 6, 8: Day 1, predose and postdose; Cycles 1 and 3: Day 1, 2 hours and 4 hours postdose; Cycles 1 and 3: Day 8, Day 15 (each cycle is 21 days)
  Time to maximum serum concentration (Tmax) will be assessed using non-compartmental methods.
Pharmacokinetic Parameter Trough Serum Concentration (Ctrough) for HER3-DXd (All Cohorts) | Cycles 1-4, 6, 8: Day 1, predose and postdose; Cycles 1 and 3: Day 1, 2 hours and 4 hours postdose; Cycles 1 and 3: Day 8, Day 15 (each cycle is 21 days)
  Trough serum concentration (Ctrough) will be assessed using non-compartmental methods.
Pharmacokinetic Parameter Area Under the Concentration Curve for HER3-DXd (All Cohorts) | Cycles 1-4, 6, 8: Day 1, predose and postdose; Cycles 1 and 3: Day 1, 2 hours and 4 hours postdose; Cycles 1 and 3: Day 8, Day 15 (each cycle is 21 days)
  Area under the concentration-time curve up to the last quantifiable time (AUClast) and Area under the concentration-time curve during dosing interval (AUCtau) will be assessed using non-compartmental methods.
Radiographic Progression-free Survival (rPFS) As Assessed by Prostate Cancer Working Group 3 (PCWG3) Criteria by the Investigator or Death Due to Any Cause Following HER3-DXd Monotherapy (Prostate Cancer Cohort Only) | From the start date of study drug to the earlier date of the first objective documentation of radiographic disease progression as assessed per PCWG3 criteria by investigator or death due to any cause, whichever occurs first, up to approximately 27 months
Proportion of Participants Achieving a ≥30% Decrease in PSA (Prostate Cancer Cohort Only) | Baseline, each cycle before infusion (each cycle is 21 days), and end of treatment, up to approximately 27 months
Time to First Subsequent Anticancer Therapy (TFST) (Prostate Cancer Cohort Only) | From the start date of study drug to initiation of the first subsequent anticancer therapy or death, whichever occurs first, up to approximately 27 months
Time to First Symptomatic Skeletal-Related Event (SSRE) (Prostate Cancer Cohort Only) | From start date of study drug to the first occurrence of any of the following: Use of EBRT, New symptomatic pathologic bone fracture, Spinal cord compression, A tumor-related orthopedic surgical intervention, up to approximately 27 months
Correlation Between HER3 Protein Expression and Efficacy | From the start date of study drug up to approximately 27 months
  HER3 protein expression in tumor tissue as determined by IHC and correlation with ORR, DoR, and PFS.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (84):
- United States (13):
  - City of Hope, Duarte, California
  - Yale Cancer Center, New Haven, Connecticut
  - AdventHealth Medical Group Oncology Research at Celebration, Kissimmee, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Health Partners Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Health Partners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - Washington University, School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute IDS, Buffalo, New York
  - Memorial Sloan Kettering Hospital, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown
  - Icon Cancer Centre Chermside, Chermside
  - Monash Medical Centre Clayton, Clayton
  - Icon Cancer Centre Hobart, Hobart
  - Icon Cancer Centre Townsville, Hyde Park
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZA, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - UZ Leuven, Leuven
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Sunnybrook Research Institute, Toronto
  - Princess Margaret Cancer Centre, Toronto
  - BC Cancer - Vancouver, Vancouver
- Sun Yat-sen University Cancer Center, Guangzhou, China
- France (9):
  - Chu Bordeaux, Bordeaux
  - Centre Georges Franăois Leclerc, Dijon
  - Hopital Claude Huriez - Chu Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hăpital de La Timone, Marseille
  - Chu Nantes - Hătel Dieu, Nantes
  - Institut Claudius Regaud, Toulouse
  - ICL - Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Krankenhaus Nordwest GmbH, Frankfurt, Germany
- Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét, Hungary
- Italy (4):
  - Humanitas Gavazzeni, Bergamo
  - IRCCS Ospedale Policlinico San Martino, Genova
  - AOU Federico II - Oncologia Clinica, Napoli
  - Centro Ricerche Cliniche di Verona s.r.l., Verona
- Japan (9):
  - Saitama Medical University International Medical Center, Hidaka
  - National Cancer Center Hospital East, Kashiwa-shi
  - NHO Shikoku Cancer Center, Matsuyama
  - Shizuoka Cancer Center, Nagaizumi-cho
  - Aichi Cancer Center Hospital, Nagoya
  - Kindai University Hospital, Osakasayama-shi
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
  - Yokohama City University Medical Center, Yokohama
- Netherlands (5):
  - Amsterdam UMC locatie Vumc, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
- Norway (3):
  - Akershus universitetssykehus, Lørenskog
  - Haukeland universitetssjukehus, Lørenskog
  - Oslo Universitetssykehus HF, Radiumhospitalet, Oslo
- South Korea (6):
  - Cha Bundang Medical Center, Cha University, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - HOSPITAL REGIONAL UNIVERSITARIO de MALAGA AVDA., Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (4):
  - University Hospital Coventry, Coventry
  - Barts Hospital, London
  - Royal Free Hospital, London
  - Nottingham City Hospital Campus, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Powles T, Bhatia A, Burtness B, Kogawa T, Nishina T, Nakayama I, Fountzilas C, Castillo DR, McKean M, Meric-Bernstam F, Colombo N, Smithy JW, Fayette J, Chandra S, Sternberg DW, Jin F, Sullivan K, Yueh S, Clinthorne G, Aguilo AE, Kudchadkar R, Hayashi H. HERTHENA-PanTumor01: a phase II study of patritumab deruxtecan (HER3-DXd) in previously treated advanced solid tumors. Future Oncol. 2025 Oct;21(25):3283-3292. doi: 10.1080/14796694.2025.2561539. Epub 2025 Oct 14. PMID 41088723